CLINICAL TRIAL: NCT00936455
Title: An Observational Study to Evaluate the Long Term Outcomes of Patients Previously Enrolled in the STRokE DOC ("STRokE DOC Trial (NCT00283868)") Telemedicine Clinical Trial.
Brief Title: Stroke Team Remote Evaluation Using a Digital Observation Camera- Long Term Outcomes(STRokE DOC-LTO)
Acronym: STRokE DOC-LTO
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brett Meyer, MD, University of California, San Diego
Other Study IDs: STRokE DOC-LTO
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Telemedicine Evaluation vs Telephone Evaluation
Keywords: telemedicine; telephone; outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Telemedicine: Telemedicine evaluated patients
- Telephone: Telephone evaluated patients

SUMMARY:
SPECIFIC AIM: The specific aims of this study are to evaluate the long term outcomes of patients previously enrolled in the STRokE DOC ("STRokE DOC Trial (NCT00283868)") telemedicine clinical trial.

AIM 1: Aim 1 is a non- randomized, retrospective, data collection study assessing long term patient outcomes of patients previously enrolled in a telemedicine vs. telephone clinical trial (STRokE DOC Trial ("STRokE DOC Trial (NCT00283868)"); now completed). STRokE DOC-LTO will evaluate, (only for those patients previously enrolled in the original telemedicine vs. telephone clinical research trial), the long term patient outcomes; comparing telemedicine versus telephone-only consultations.

DETAILED DESCRIPTION:
SPECIFIC AIM: The specific aims of this study are to evaluate the long term outcomes of patients previously enrolled in the STRokE DOC ("STRokE DOC Trial (NCT00283868)") telemedicine clinical trial.

AIM 1: Aim 1 is a non- randomized, retrospective, data collection study assessing long term patient outcomes of patients previously enrolled in a telemedicine vs. telephone clinical trial (STRokE DOC Trial ("STRokE DOC Trial (NCT00283868)"); now completed). STRokE DOC-LTO will evaluate, (only for those patients previously enrolled in the original telemedicine vs. telephone clinical research trial), the long term patient outcomes; comparing telemedicine versus telephone-only consultations.

Specific Protocol Information: The protocol will contact these patients by telephone. One of 5 Stroke Center team members will contact the patient, using strict telephone scripted language (approved by the IRB) and ask questions regarding

1. current functional status
2. death
3. Hemorrhage
4. Recurrent Stroke
5. Disposition for 3 time periods (6 months after index event, 12 months after index event, and "current" time of contact.

ELIGIBILITY:
Inclusion Criteria are:

1. Male or female subjects, age > 18 years.
2. Prior enrollment into the STRokE DOC ("STRokE DOC Trial (NCT00283868)") clinical research trial.

Exclusion criteria are:

1. Male or female subjects, age < 18 years.
2. Patients not previously enrolled into the STRokE DOC ("STRokE DOC Trial (NCT00283868)") clinical research trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria are:
  1. Male or female subjects, age > 18 years.
  2. Prior enrollment into the STRokE DOC ("STRokE DOC Trial (NCT00283868)") clinical research trial.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett C Meyer, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD, San Diego, California, United States

REFERENCES:
- [Background] Meyer BC, Raman R, Hemmen T, Obler R, Zivin JA, Rao R, Thomas RG, Lyden PD. Efficacy of site-independent telemedicine in the STRokE DOC trial: a randomised, blinded, prospective study. Lancet Neurol. 2008 Sep;7(9):787-95. doi: 10.1016/S1474-4422(08)70171-6. PMID 18676180
- [Derived] Meyer BC, Raman R, Ernstrom K, Tafreshi GM, Huisa B, Stemer AB, Hemmen TM. Assessment of long-term outcomes for the STRokE DOC telemedicine trial. J Stroke Cerebrovasc Dis. 2012 May;21(4):259-64. doi: 10.1016/j.jstrokecerebrovasdis.2010.08.004. Epub 2010 Sep 19. PMID 20851629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were assessed in July 2009. Patients were all contacted at a single time point (irrespective of time since original trial enrollment) and were asked structured questions regarding their level of function at 3 time points (6 months after original event, 12 months after original event, and current time point).
Pre-assignment Details: Observational study. Patient contact via telephone. Patients were all contacted at a single time point (irrespective of time since original trial enrollment) and were asked structured questions regarding their level of function at 3 time points (6 months after original event, 12 months after original event, and current time point).
Groups:
- Telemedicine: Telemedicine evaluated patients- The definition of telemedicine for this trial was the use of 2 way video and 2 way audio videoconferencing and also the use of digital access to radiology image review. Telephone use is not considered telemedicine for the purposes of this trial.
Period: Overall Study
Arm/Group | Telemedicine | Telephone
Started | 37 | 38
Completed | 37 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telemedicine | Telephone | Total
Number analyzed (Participants) | 37 | 38 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (13) | 67 (13) | 67 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 19 | 22 | 41
Region of Enrollment [Number; unit: participants]
  United States | 37 | 38 | 75

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome (mRS(0-1)) at 6 Months After Index Event. The mRS is the Modified Rankin Scale That Measures Patient's Functional Level of Activity. The Scale is a 6 Point Scale With 0 Score Being Normal and 6 Score Being Death.
Description: Functional Outcome (mRS(0-1)) at 6 months after index event. The mRS is the modified Rankin Scale that measures patient's functional level of activity. The scale is a 6 point scale with 0 score being normal and 6 score being death. Listed below is the number of participants in each group with Functional Outcome (mRS(0-1)).
Time Frame: Patients were all assessed at a single time point (July 2009) for retrospective reporting of how they were at 6 months since initial event (Primary endpoint). The average time per participant relative to the study entry time in concrete units is 6 months
Population: NUMBER OF PARTICIPANTS WAS DETERMINED BASED ON PER PROTOCOL NUMBER OF PATIENT ABLE TO BE CONTACTED VIA TELEPHONE
Measure: Number; unit: participants
Groups:
- Telemedicine: Functional Outcome (mRS(0-1)) at 6 months after index event in the telemedicine group
- Telephone: Functional Outcome (mRS(0-1)) at 6 months after index event in the telephone group
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 37 | 38
participants | 12 | 17

2. Secondary Outcome: Recurrent Stroke
Description: Assessing amount of patients that had recurrent stroke by 6 months (patients that retrospectively reporting having had a stroke from 0-6 months after their index event)
Time Frame: as for outcome 1
Population: NUMBER OF PARTICIPANTS WAS DETERMINED BASED ON PER PROTOCOL NUMBER OF PATIENT ABLE TO BE CONTACTED VIA TELEPHONE
Measure: Number; unit: participants
Groups:
- Telemedicine: Assessing amount of patients that had recurrent stroke by 6 months (patients that retrospectively reporting having had a stroke from 0-6 months after their index event)
- Telephone: Recurrent stroke at 6 months in each group
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 37 | 38
participants | 1 | 2

3. Secondary Outcome: Recurrent Stroke
Description: Assessing amount of patients that had recurrent stroke by 12 months (patients that retrospectively reporting having had a stroke from 6-12 months after their index event)
Time Frame: Patients were all assessed at a single time point (July 2009) for retrospective reporting of how they were at 12 months since initial event (2ndary endpoint). The average time per participant relative to the study entry time in units is 12 months
Population: NUMBER OF PARTICIPANTS WAS DETERMINED BASED ON PER PROTOCOL NUMBER OF PATIENT ABLE TO BE CONTACTED VIA TELEPHONE
Measure: Number; unit: participants
Groups:
- Telemedicine: Assessing amount of patients that had recurrent stroke by 12 months (patients that retrospectively reporting having had a stroke from 6-12 months after their index event)
- Telephone: Assessing number of recurrent strokes by 12 months
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 37 | 38
participants | 0 | 1

4. Secondary Outcome: Functional Outcome (mRS(0-1)) at 12 Months After Index Event. The mRS is the Modified Rankin Scale That Measures Patient's Functional Level of Activity. The Scale is a 6 Point Scale With 0 Score Being Normal and 6 Score Being Death.
Description: Functional Outcome (mRS(0-1)) at 12 months after index event. The mRS is the modified Rankin Scale that measures patient's functional level of activity. The scale is a 6 point scale with 0 score being normal and 6 score being death. Listed below is the number of participants in each group with Functional Outcome (mRS(0-1)).
Time Frame: as for outcome 3
Population: NUMBER OF PARTICIPANTS WAS DETERMINED BASED ON PER PROTOCOL NUMBER OF PATIENT ABLE TO BE CONTACTED VIA TELEPHONE
Measure: Number; unit: participants
Groups:
- Telemedicine: Functional Outcome (mRS(0-1)) at 12 months after index event in telemedicine group
- Telephone: Functional Outcome (mRS(0-1)) at 12 months after index event in telephone group
Arm/Group | Telemedicine | Telephone
Number analyzed (Participants) | 37 | 38
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Observational Trial- Adverse events were not collected/ assessed in this observational study
Description: Observational Trial- Adverse events were not collected/ assessed in this observational study
Arm/Group | Telemedicine | Telephone
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This is an observational trial where patients were contacted by telephone for data collection only. No adverse event information was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No